CLINICAL TRIAL: NCT04779515
Title: Effect of Low-pressure Pneumoperitoneum on Pain and Inflammation Post Laparoscopic Cholecystectomy: A Randomized, Double-blinded, Controlled, Clinical Trial.
Brief Title: Effect of Low-pressure Pneumoperitoneum on Pain and Inflammation Post Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Ibrahim Mansour, Dr. Hanan Mansour, post-graduate, general surgery resident, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2243
Record Dates: First submitted 2021-02-27; First posted 2021-03-03 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Pneumoperitoneum; Pain; Inflammation
Keywords: low-pressure pneumoperitoneum, lap chole
MeSH Terms: conditions — Pneumoperitoneum; Pain; Inflammation

STUDY DESIGN:
Intervention Model Description: participants were divided into two masked groups, labelled red and green; those operated at low-pressure pneumoperitoneum (green-label) and those operated at standard-pressure pneumoperitoneum (red-label).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: none of the participants knew at which pressure they will be operated on, nor the physicians who followed participants at floor or those analyzing blood samples, not the assigned physician to collect data, nor the personnel doing the analysis.
  only the operating surgeon and circulating nurse were aware of the meaning of the participant assigned label at time of operation. The masking was revealed post completion of analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-pressure (Experimental): Participants undergone laparoscopic cholecystectomy by creation of a low-pressure pneumoperitoneum, set at 8-10 mm Hg
  Interventions: Procedure: low-pressure pneumoperitoneum
- Standard-pressure (Active Comparator): Participants undergone laparoscopic cholecystectomy by creation of a standard-pressure pneumoperitoneum, set at 12-14 mm Hg
  Interventions: Procedure: standard-pressure pneumoperitoneum

INTERVENTIONS:
Procedure: low-pressure pneumoperitoneum — insufflation of the abdomen for creation of pneumoperitoneum, pressure set points between 8 to 10 mm Hg
  Arms: Low-pressure
Procedure: standard-pressure pneumoperitoneum — insufflation of the abdomen for creation of pneumoperitoneum, pressure set points between 12 to 14 mm Hg
  Arms: Standard-pressure

SUMMARY:
The purpose of this study is to assess the effect of low-pressure pneumoperitoneum on post operative pain and inflammation in patients undergoing elective laparoscopic cholecystectomy by comparing it to standard practice.

DETAILED DESCRIPTION:
After obtaining informed consent from eligible study participants. patients were randomized into one of two masked groups, labelled red and green. The red-label group was operated at standard-pressure pneumoperitoneum, while the green-label group was operated at low-pressure pneumoperitoneum. Baseline blood samples were obtained pre-operatively for ten inflammatory markers, patients' demographics and intra-operative details collected, then post-operative pain and change in inflammatory markers were followed.

ELIGIBILITY:
Inclusion Criteria:

* Elective admission for laparoscopic cholecystectomy

Exclusion Criteria:

* Current or previous diagnosis of acute cholecystitis confirmed by ultrasound
* previous GI surgeries, except bariatric and anti-reflux surgeries
* Currently on immunosuppressant agents
* Pregnancy
* Breastfeeding
* Currently diagnosed with drug addiction
* American Society of Anesthesiologists (ASA) score 3 and more

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
change from baseline in pain on the 11-point short pain scale (SPS-11) at hour 12 post-op | baseline and 12 hours post-op
  the SPS-11 is a validated, self-reported numeric instrument assessing pain intensity, ranging from 0 to 10; where 0 is no pain, and 10 is the worst pain felt ever.
  change = (pain score at 12-hr post-op) - (baseline pain score assessed at 6-hr post-op)
change from baseline in pain on the 11-point short pain scale (SPS-11) at hour 24 post-op | baseline and 24 hours post-op
  the SPS-11 is a validated, self-reported numeric instrument assessing pain intensity, ranging from 0 to 10; where 0 is no pain, and 10 is the worst pain felt ever.
  change = (pain score at 24-hr post-op) - (baseline pain score assessed at 6-hr post-op)
change from baseline in pain on the 11-point short pain scale (SPS-11) at day 7 post-op | baseline and 7 days post-op
  the SPS-11 is a validated, self-reported numeric instrument assessing pain intensity, ranging from 0 to 10; where 0 is no pain, and 10 is the worst pain felt ever.
  change = (pain score at post-op day 7) - (baseline pain score assessed at 6-hr post-op)
change from baseline in WBC count at 24hr post op | baseline and 24 hours post-op
  calculate the rise in white blood cycles count as inflammatory marker post-op in 1000 cells per cubic millimeter of blood.
  change = (post-op WBC count) - (baseline WBC count)
change from baseline in Plt count at 24hr post op | baseline and 24 hours post-op
  calculate the rise in platelets count as inflammatory marker post-op in × 10^9/L of blood change = (post-op Plt count) - (baseline Plt count)
change from baseline in ESR value at 24hr post op | baseline and 24 hours post-op
  calculate the rise in erythrocyte sedimentation rate value as inflammatory marker post-op in millimeters per hour.
  change = (post-op ESR) - (baseline ESR)
change from baseline in CRP level at 24hr post op | baseline and 24 hours post-op
  calculate the rise in C reactive protein level as inflammatory marker post-op in mg/L change = (post-op CRP) - (baseline CRP)
change from baseline in Alb level at 24hr post op | baseline and 24 hours post-op
  calculate the drop in albumin level as inflammatory marker post-op in g/dL change = (baseline Alb) - (post-op baseline Alb)
change from baseline in cortisol level at 4hr post op | baseline and 4 hours post-op
  calculate the rise in cortisol level as inflammatory marker post-op in nmol/L change = (post-op cortisol ) - (baseline cortisol )
change from baseline in IL-6 level at 24hr post op | baseline and 24 hours post-op
  calculate the rise in interleukin 6 level as inflammatory marker post-op in pg/mL change = (post-op IL-6) - (baseline IL-6)
change from baseline in IL-17 level at 24hr post op | baseline and 24 hours post-op
  calculate the rise in interleukin 17 level as inflammatory marker post-op in pg/mL change = (post-op IL-17) - (baseline IL-17)
change from baseline in IL-1 level at 24hr post op | baseline and 24 hours post-op
  calculate the rise in interleukin 1 level as inflammatory marker post-op in pg/mL change = (post-op IL-1) - (baseline IL-1)
change from baseline in TNF level at 24hr post op | baseline and 24 hours post-op
  calculate the rise in tumor necrosis factor alpha level as inflammatory marker post-op in pg/mL change = (post-op TNF) - (baseline TNF)

SECONDARY OUTCOMES:
Difference in surgery difficulty level among two groups | through study completion, an average of 1 year
  assessing level of surgery difficulty between low and standard pressure pneumoperitoneum groups.
  Difficulty was self reported by operating surgeon as easy (score=1), moderate (score=2), or difficult (score=3).
  Difference assessed by calculating average between groups
Difference in surgery time among two groups | through study completion, an average of 1 year
  assessing difference in insufflation time calculated in minutes between low and standard pressure pneumoperitoneum groups.
  insufflation time was calculated from time of creation of pneumoperitoneum to deflation of the abdomen.
  Difference assessed by calculating average between groups

CONTACTS AND LOCATIONS:
Overall Officials: Salam Daradkeh, Prof., Study Chair — University of Jordan; Mohammad Rashdan, Prof., Principal Investigator — University of Jordan; Raed Al-Taher, Prof., Study Director — University of Jordan
Locations (1):
- Jordan University Hospital, Amman, Jubaiha, Jordan

IPD SHARING:
Plan to Share IPD: Yes
we are willing to share all study data for interested researchers to conduct secondary studies of their own.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the data will be available from April,2021 up to the end of 2021 year
Access Criteria: Data will be shared for medical investigators interested in the topic of pneumoperitoneum, to request please contact (hanan.ju@gmail.com)